CLINICAL TRIAL: NCT06666712
Title: Chronic Convection Enhanced Delivery of Topotecan for Recurrent Malignant Glioma
Brief Title: Chronic CED of TPT for Recurrent Malignant Glioma
Acronym: TPT CED rHGG
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jeffrey N. Bruce (Other)
Responsible Party: Sponsor-Investigator, Jeffrey N. Bruce, Professor of Neurological Surgery, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAV1710
Record Dates: First submitted 2024-10-05; First posted 2024-10-31 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Brain Tumor, Recurrent; Malignant Glioma (WHO Grade III or IV); IDH1/IDH2 Mutation
Keywords: Brain Tumors; topotecan; Convection-Enhanced Delivery (CED); Glioma; IDH Mutation
MeSH Terms: conditions — Brain Neoplasms; Glioma; Lymphoma, Follicular | interventions — Topotecan; 9 alpha,11 alpha,15 alpha-trihydroxy-16-phenoxy-17,18,19,20-tetranorprosta-4,5,13-trienoic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Long-term CED of Topotecan (Experimental): Six patients will be treated with Topotecan by Convection-Enhanced Delivery. Four 48-hour Topotecan infusions will be carried out over the course of 23-29 days (with five to seven-day drug holiday after the first three infusions). Infusions will take place using Synchromed II infusion pumps with the same infusion parameters and experimental conditions used in our previous Phase I clinical trial and other short-term studies.
  Interventions: Drug: Topotecan

INTERVENTIONS:
Drug: Topotecan — Topotecan (TPT) is a chemotherapeutic agent that is a topoisomerase inhibitor. This intervention is uniquely distinguished through its administration using an externalized catheter and external microinfusion pump (Convection-Enhanced Delivery)
  Other Names: TPT; Hycamtin

SUMMARY:
The primary goal of this study is to establish the safety of chronic Convection Enhanced Delivery (CED) of the chemotherapeutic drug Topotecan for patients with recurrent malignant glioma that harbors the Isocitrate Dehydrogenase mutation (IDH-mut). The secondary goal of the study is to study drug distribution and assess the tumor response to prolonged continuous CED of Topotecan.

Convection Enhanced Delivery is a novel method of drug delivery that allows administration of a drug directly to the brain. In CED, a drug pump is placed under the skin in the chest or abdominal region. The pump is connected to a catheter that is tunneled underneath the skin to the brain. The tip of the catheter then infuses Topotecan directly onto the brain tumor. There will be a total of four treatment infusions over the course of 23-29 days, with a 5-7-day rest period between each infusion. Throughout this period, patients' health will be monitored through imaging, blood draws, and regular exams. At the end of the treatment period, the pump will be removed, followed by resection of the tumor. Patients will be followed for the duration of their lives.

This is the investigator's second clinical trial studying CED of TPT in recurrent glioma. In the prior Phase 1b trial, chronic pulsatile CED safely and effectively delivered Topotecan to patients with IDH mutant recurrent Glioblastoma (WHO grade 4).

DETAILED DESCRIPTION:
Malignant gliomas are among the most pernicious of human tumors. They are locally invasive and universally recurrent, often recurring within two centimeters of the original resection cavity. Although numerous chemotherapeutic drugs demonstrate significant anti-tumor activity in preclinical studies, their efficacy in clinical trials has been dismal; systemic delivery fails to achieve therapeutic drug levels in tumor cells due to various factors including limited blood-brain barrier permeability and systemic toxicity.

Convection-Enhanced Delivery (CED) can circumvent this challenge by delivering therapeutics directly to the brain, bypassing systemic circulation and the blood-brain barrier. CED uses a subcutaneously implanted catheter-pump system, enabling sustained, prolonged delivery while foregoing the need for an external catheter and bedside pump. In the most recent Phase Ib clinical trial, chronic pulsatile CED safely and effectively delivered Topotecan (TPT), a topoisomerase I inhibitor, to patients with recurrent Glioblastoma (WHO grade 4), Isocitrate Dehydrogenase wild type (IDH-WT). However, malignant glioma displays marked genetic and phenotypic heterogeneity not fully reflected by IDH-WT glioblastoma. In the current study, the investigators aim to further demonstrate the safety and efficacy of this drug delivery system in IDH mutated malignant glioma. The investigators hypothesize that extended chronic pulsatile local-regional delivery of TPT continues to be safe, effective, and feasible in patients with recurrent IDH mutated WHO grade 3-4 malignant glioma. This study will use the previously established method of CED through subcutaneously implanted pumps combined with non-invasive imaging to monitor drug distribution. As in the previous study, the drug's distribution will be characterized using an innovative, non-invasive methodology for measuring intracerebral distribution.

The hypothesis is that intracerebral CED can safely, effectively, and chronically administer TPT to patients with recurrent malignant glioma, including WHO grade 3-4 IDH1/2 mutated subtypes, and drug distribution can be measured non-invasively. The inclusion of IDH1/2 mutated glioma (WHO grade 3-4) marks an expansion from our prior Phase Ib trial to better reflect the heterogeneity of malignant glioma.

The chronic CED and non-invasive imaging methodology was developed in the porcine model and was subsequently shown to be safe for patients with recurrent WHO grade 4 glioma in the phase Ib clinical trial. Similar to the previous trial design, patients will undergo implantation of the CED catheters and subcutaneously implanted pumps, after which four cycles of TPT/gadolinium will be administered. Each cycle will include 48 hours of active drug infusion followed by five to seven days of drug holiday. Following the four cycles, the catheters and pumps will be removed and tumors will be resected. Tumoral and parenchymal distribution of gadolinium (measured by MRI) will be correlated with TPT levels (measured by mass spectrophotometry) in tissue samples obtained upon tumor resection. Cytotoxic response to TPT will be investigated by both MRI and direct histologic comparison between tissue samples taken at resection versus initial biopsy and MRI.

At the conclusion of these studies, the investigators expect to demonstrate the safe and successful delivery of chronic, high doses of TPT directly into patients' tumors, thereby avoiding the limitations imposed by conventional systemic delivery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have recurrent malignant glioma with a history of WHO grade 3-4 IDH-mutant status and evidence of radiographic progression and suspicion of histopathological recurrence. Stereotactic biopsies will be performed to assess the presence of active tumor by frozen section prior to initiating treatment. Patients with a history of WHO grade 2 recurrent glioma, IDH-Mutant, who now demonstrate high-grade features of IDH-mutant WHO grade 3-4 will also be included.
2. Patients with recurrent malignant glioma, IDH-mutant, who have failed standard of care treatment are eligible.
3. An MRI scan must be obtained within 30 days of enrollment and must demonstrate an enhancing mass without significant mass effect. Tumors must be less than 32 cc in total volume as assessed by the principal investigator based on pre-enrollment MRI. The lesion must be stereotactically accessible.
4. Karnofsky performance score must be greater than or equal to 70.
5. Men and women of childbearing potential must practice birth control. Women of childbearing potential must have a urine pregnancy test within 7 days of study entry. In accordance with topotecan administration guidelines, women must practice birth control for at least 1 month following chemotherapy infusion. Men must practice birth control for at least four months following termination of chemotherapy infusion.
6. Patients or appropriate legally authorized representatives must possess the ability to give Informed Consent.
7. Patients must be willing to and medically capable of undergoing the surgical operation.
8. Patients must be at least 18 years old.
9. Patients must not have known abnormal organ and marrow function as defined below 14 days or fewer from registration:

   * Leukocytes: ≥3,000/mcL
   * Absolute neutrophil count : ≥1,500/mcL
   * Platelets: ≥100,000/mcL
   * Total bilirubin: within normal institutional limits
   * AST(SGOT)/ALT(SGPT): ≤2.5 × institutional upper limit of normal
   * Creatinine: within normal institutional limits OR
   * Creatinine clearance: ≥60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.

Exclusion Criteria:

1. Patients with diffuse subependymal or CSF disease.
2. Patients with tumors involving the cerebellum or both cerebral hemispheres.
3. Patients with an active infection requiring treatment or having an unexplained febrile illness.
4. Patients who are known HIV, Hepatitis B or Hepatitis C positive. HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with Topotecan. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated. HIV, Hepatitis B and Hepatitis C testing is not required for patients not known to have these infections.
5. Patients with systemic diseases which may be associated with unacceptable anesthetic/operative risk.
6. Patients who have previously received systemic topotecan for their tumor.
7. Patients who are not able to receive MRI or PET scans.
8. History of allergic reactions attributed to compounds of similar chemical or biologic composition to topotecan, other topoisomerase inhibitors or gadolinium compounds.
9. Patients who are currently receiving treatment with agents that are metabolized solely through cytochrome P450 (CYP) 3A4/5 (CYP3A4/5) and have a narrow therapeutic index or are strong CYP2C8 inhibitors. Patients who are receiving treatment with agents that carry a risk for QT prolongation and are CYP3A substrates are also ineligible. Caution should be used in patients taking other CYP2C8 - or CYP3A4/5-interacting agents as they may increase the serum concentrations of topotecan. If previously on such agents, the patient must discontinue them for at least two weeks prior to study treatment.
10. Patients with uncontrolled intercurrent illness including, but not limited to, ongoing active infection, systemic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
11. Women of childbearing potential who fail to demonstrate a negative pregnancy test 7 or fewer days from registration.
12. Women who are breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Safety, defined as dose at which all patients have had no greater than grade 2 adverse reactions | Up to 29 days
  The primary outcome of the study is to measure the safety of prolonged CED of Topotecan in patients with recurrent IDH-mutant malignant glioma. Safety is defined as the dose at which all patients have had no greater than grade 2 adverse reactions possibly, probably, or definitely related to CED of Topotecan as measured through physical and neurologic examination, laboratory studies, radiographic studies, and adverse effects, as defined by the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 out from Grade 1 (mild symptoms) to Grade 5 (death related to adverse event).

SECONDARY OUTCOMES:
Progression Free Survival (PFS), Overall Survival (OS) | Up to 5 years
  Progression Free Survival is defined as the duration of time from start of Topotecan treatment to time of progression or death from any cause, whichever occurs first. Overall survival is defined as the duration of time from the start of Topotecan treatment to death from any cause. Patients will be contacted every 3-6 months, up to 5 years, by phone until death.
Tumor Response to Treatment | Up to 29 days of treatment, and 4-6 weeks post treatment period
  The response of the tumor to TPT treatment will be measured radiographically with MRI periodically throughout the 23-29 day treatment period and on follow up 4-6 weeks after treatment, per the international criteria proposed by the updated Response Assessment in Neuro-oncology (RANO) guidelines.
Clinical Toxicity Rate | Up to 29 days
  This is defined by the number of serious adverse events occuring, which is projected to be ≤ 5% at 23-29 days. A clinical toxicity rate that exceeds 20% will be considered unacceptable for this procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Bruce, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center / NewYork-Presbyterian Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sonabend AM, Stuart RM, Yun J, Yanagihara T, Mohajed H, Dashnaw S, Bruce SS, Brown T, Romanov A, Sebastian M, Arias-Mendoza F, Bagiella E, Canoll P, Bruce JN. Prolonged intracerebral convection-enhanced delivery of topotecan with a subcutaneously implantable infusion pump. Neuro Oncol. 2011 Aug;13(8):886-93. doi: 10.1093/neuonc/nor051. Epub 2011 Jul 12. PMID 21750007
- [Background] Yan H, Parsons DW, Jin G, McLendon R, Rasheed BA, Yuan W, Kos I, Batinic-Haberle I, Jones S, Riggins GJ, Friedman H, Friedman A, Reardon D, Herndon J, Kinzler KW, Velculescu VE, Vogelstein B, Bigner DD. IDH1 and IDH2 mutations in gliomas. N Engl J Med. 2009 Feb 19;360(8):765-73. doi: 10.1056/NEJMoa0808710. PMID 19228619
- [Background] Han S, Liu Y, Cai SJ, Qian M, Ding J, Larion M, Gilbert MR, Yang C. IDH mutation in glioma: molecular mechanisms and potential therapeutic targets. Br J Cancer. 2020 May;122(11):1580-1589. doi: 10.1038/s41416-020-0814-x. Epub 2020 Apr 15. PMID 32291392
- [Background] Spinazzi EF, Argenziano MG, Upadhyayula PS, Banu MA, Neira JA, Higgins DMO, Wu PB, Pereira B, Mahajan A, Humala N, Al-Dalahmah O, Zhao W, Save AV, Gill BJA, Boyett DM, Marie T, Furnari JL, Sudhakar TD, Stopka SA, Regan MS, Catania V, Good L, Zacharoulis S, Behl M, Petridis P, Jambawalikar S, Mintz A, Lignelli A, Agar NYR, Sims PA, Welch MR, Lassman AB, Iwamoto FM, D'Amico RS, Grinband J, Canoll P, Bruce JN. Chronic convection-enhanced delivery of topotecan for patients with recurrent glioblastoma: a first-in-patient, single-centre, single-arm, phase 1b trial. Lancet Oncol. 2022 Nov;23(11):1409-1418. doi: 10.1016/S1470-2045(22)00599-X. Epub 2022 Oct 13. PMID 36243020
- [Background] Bruce JN, Fine RL, Canoll P, Yun J, Kennedy BC, Rosenfeld SS, Sands SA, Surapaneni K, Lai R, Yanes CL, Bagiella E, DeLaPaz RL. Regression of recurrent malignant gliomas with convection-enhanced delivery of topotecan. Neurosurgery. 2011 Dec;69(6):1272-9; discussion 1279-80. doi: 10.1227/NEU.0b013e3182233e24. PMID 21562434
- [Background] Bhowmik A, Khan R, Ghosh MK. Blood brain barrier: a challenge for effectual therapy of brain tumors. Biomed Res Int. 2015;2015:320941. doi: 10.1155/2015/320941. Epub 2015 Mar 19. PMID 25866775